CLINICAL TRIAL: NCT00965952
Title: A Prospective, Observational Surgical Simulation Study to Evaluate the Safety of the VFIX Device Mechanism as Treatment for Vaginal Apical Prolapse
Brief Title: A Surgical Simulation Study to Evaluate the Safety of a Device Mechanism as Treatment for Vaginal Apical Prolapse
Status: Completed | Type: Observational
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: David Robinson MD/Medical Director, Ethicon
Other Study IDs: 300-08-009
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this pilot study is to perform a procedure to evaluate the safety of the placement of a new device (known as the VFIX device).

DETAILED DESCRIPTION:
In this study, the surgeon will not use the actual V-Fix device. Instead, the surgeon will use a routine operating room instrument, which is similar to the size and shape of the V-Fix device to mimic the placement of the VFIX device by using the routine operating room instrument to push the top of your vagina towards the ligament.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Subjects with apical support prolapse in whom the surgeon may consider a surgical procedure to correct level 1 support, with "C" or "D" descent at least halfway down the vaginal length (i.e. uterus and cervix or the vaginal vault in hysterectomised subjects), and having laparoscopy or abdominal surgery (additional surgery e.g. tubal ligation or ovarian cystectomy is also allowed).
* Vaginal examination during the screening visit confirms that the lateral fornix of the vagina can reach both the left and right SSL and therefore the surgical simulation can be performed.
* The investigator considers that the subject is medically fit enough to receive extended anaesthesia of approximately 15 minutes, to complete the additional anatomical observation study procedures.
* Subjects agree to participate in the study and document this agreement by signing the Ethics Committee approved informed consent.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital referrals
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Incidence of subjects without any bowel entrapment between the vagina and the right SSL in subjects that the surgeon declares he would have deployed the V-Fix device | Intraoperative

SECONDARY OUTCOMES:
Incidence of subjects without any bladder entrapment or traversing of the peritoneal cavity between the vagina and the right or left SSL in subjects that the surgeon declares he would have deployed the V-Fix device | Intraoperative
Incidence of subjects without any bowel entrapment between the vagina and the left SSL in subjects that the surgeon declares he would have deployed the V-Fix device | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: David Robinson, MD, Study Director — Ethicon, Inc.
Locations (4):
- Australia (4):
  - North Shore Private Hospital, Sydney, New South Wales
  - St George Private Hospital, Sydney, New South Wales
  - Frances Perry House, Melbourne, Victoria
  - Royal Women's Hospital, Melbourne, Victoria